CLINICAL TRIAL: NCT06970301
Title: A Single-center, Placebo-controlled, Participant-blind, Investigator-blind, Randomized, Multiple Ascending Dose in Titration Study to Assess The Safety and Tolerability, and Pharmacokinetics of UCB0022 in Healthy Caucasian, Japanese, and Chinese Participants
Brief Title: A Study to Assess the Safety and Tolerability, and Pharmacokinetics of UCB0022 in Healthy Caucasian, Japanese, and Chinese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0135
Record Dates: First submitted 2025-05-12; First posted 2025-05-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy Study Participants
Keywords: Healthy Study Participants; Phase 1; ascending dose; UCB0022; glovadalen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a participant- and investigator-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Caucasian) (Experimental): Study participants randomized to Cohort 1 (Part A) will receive multiple ascending doses of glovadalen or matching placebo (PBO) at pre-specified time points during the Treatment Period.
  Interventions: Drug: glovadalen; Other: Placebo
- Cohort 2 (Japanese) (Experimental): Study participants randomized to Cohort 2 (Part B) will receive multiple ascending doses of glovadalen or matching PBO at pre-specified time points during the Treatment Period.
  Interventions: Drug: glovadalen; Other: Placebo
- Cohort 3 (Chinese) (Experimental): Study participants randomized to Cohort 3 (Part B) will receive multiple ascending doses of glovadalen or matching PBO at pre-specified time points during the Treatment Period.
  Interventions: Drug: glovadalen; Other: Placebo

INTERVENTIONS:
Drug: glovadalen — Study participants will receive doses of glovadalen (UCB0022) at pre-specified time points during the Treatment Period of Part A and Part B.
  Other Names: UCB0022
Other: Placebo — Study participants will receive matching placebo at pre-specified time points during the Treatment Period of Part A and Part B.
  Other Names: PBO

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of oral glovadalen (UCB0022) in healthy Caucasian, Japanese, and Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF).
* Participants who are overtly healthy (in the opinion of the investigator) as determined by medical evaluation including medical history (any chronic and acute illness), physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory tests during the Screening Period. Participants with test results that are outside the specified normal ranges and that are deemed not clinically significant will be allowed at the discretion of the investigator. If participants have a test result outside the specific range that is deemed clinically significant, repeat of the investigation may be allowed at the discretion of the investigator.
* For Japanese participants: Participants are of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (participant have all 4 Japanese grandparents born in Japan) and have not had a significant change in lifestyle or diet since leaving Japan.
* For Chinese participants: Participants are of Chinese descent as evidenced by appearance and verbal confirmation of familial heritage (a participant has all 4 Chinese grandparents born in China) and have not had a significant change in lifestyle or diet since leaving China.
* For Caucasian participants: Participants are of Caucasian descent as evidenced by appearance and verbal confirmation of familial heritage with all 4 grandparents of Caucasian descent.

Weight

- Participants with body weight ≥45 kilogram (kg) and body mass index (BMI) within the range of 18.0 to 30.0 kg/m^2 (inclusive).

Sex and contraceptive/barrier requirements

* Male and female

  1. Male participants must agree to use contraception of the full protocol during the Treatment Period and for 14 days after the final dose of study intervention and refrain from donating sperm during this period.
  2. Female participants are eligible to participate if they are not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

     Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance of the full protocol during the Treatment Period and for at least 14 days after the final dose of study intervention

     Exclusion Criteria:
* Participants have any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the participants' ability to participate in this study.
* Participants have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, cerebrovascular, neurological, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data in the opinion of the investigator.
* History of hypertension, hypertensive crisis, hypertensive encephalopathy, or orthostatic hypotension, unless the underlying cause was unequivocally identified and has been removed.
* History of ischemic stroke, transient ischemic attack, angina, myocardial infarction, any systemic embolism, any clinically significant arrythmia, or congestive heart failure
* Participants have the following liver enzyme test results during the Screening Period or Day -1:

  1. aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN), (isolated bilirubin <1.5xULN is acceptable if fractionated and direct bilirubin <35%).
  2. Tests that result in ALT, AST, bilirubin, or ALP up to 25% above the exclusion limit may be repeated once for confirmation.
* Participants have current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones).
* Participants have 12-lead ECG with changes considered to be clinically significant (eg, QTcF >450 ms in males and >470 ms in females based on average of triplicate ECGs, left bundle branch block, evidence of myocardial ischemia, or second-degree Type II atrioventricular block) during the Screening Period or Day -1.
* Participants have a history of risk factors for torsades de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
* Participants have had any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Participants have had breast cancer within the past 10 years.
* Participants have a history of a major organ transplant or hematopoietic stem cell/marrow transplant.
* Participants have a current history of alcohol or drug use disorder, as defined in Diagnostic and Statistical Manual of Mental Disorders Version 5, within the last year.
* Participants have a known hypersensitivity to any components of the study intervention as stated in the protocol.
* Participants have a history of severe allergic reaction that required medical intervention.
* Participants have clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnea, sore throat, fatigue, anosmia, ageusia) or had a positive SARS CoV 2 test result within the last 4 weeks prior to dosing.
* Active treatment or a history of glaucoma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Occurrence of TEAEs (Part A) | From Baseline to the end of Safety Follow-up Period (up to 49 days)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) are adverse events not present prior to the pharmaceutical product administration or an already present event that worsens either in intensity or frequency.
Occurrence of TEAEs (Part B) | From Baseline to the end of Safety Follow-up Period (up to 44 days)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) are adverse events not present prior to the pharmaceutical product administration or an already present event that worsens either in intensity or frequency.

SECONDARY OUTCOMES:
Cmax (Part A) | Day 1 in Part A
  Cmax: maximum observed plasma concentration
Cmax,ss (Part A) | From Day 10 to Day 37 in Part A
  Cmax: maximum observed plasma concentration at steady state condition
AUC0-24 (Part A) | Day 1 in Part A
  AUC0-24: area under the plasma concentration-time curve from time zero to 24 hours
AUC0-24,ss (Part A) | From Day 10 to Day 37 in Part A
  AUC0-24,ss: area under the plasma concentration-time curve from time zero to 24 hours at steady state condition
AUC0-t (Part A) | Day 1 in Part A
  AUC0-t: area under the plasma concentration-time curve from time zero to the last quantifiable concentration
AUC0-t,ss (Part A) | From Day 10 to Day 37 in Part A
  AUC0-t,ss: area under the plasma concentration-time curve from time zero to the last quantifiable concentration at steady state condition
Cmax (Part B) | Day 1 in Part B
  Cmax: maximum observed plasma concentration
Cmax,ss (Part B) | From Day 5 to Day 32 in Part B
  Cmax: maximum observed plasma concentration at steady state condition
AUC0-24 (Part B) | Day 1 in Part B
  AUC0-24: area under the plasma concentration-time curve from time zero to 24 hours
AUC0-24,ss (Part B) | From Day 5 to Day 32 in Part B
  AUC0-24,ss: area under the plasma concentration-time curve from time zero to 24 hours at steady state condition

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- Up0135 1001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual patient-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.